CLINICAL TRIAL: NCT06391047
Title: The Impact of Mulligan Squeeze Technique as an Adjunct to Conventional Physiotherapy on Meniscal Derangement in Knee Osteoarthritis Patients
Brief Title: Impact of Mulligan Squeeze Technique on Meniscal Derangement in Knee Osteoarthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Dr Izza Ayub; PT, Dr Izza Ayub;PT Lecturer, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TUF/DR/SA/MSPP/2024/383
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis, Knee; Knee Injuries; Meniscus; Derangement; Meniscus Tear; Meniscus Lesion
Keywords: Knee Osteoarthritis; manual therapy intervention; rehabilitation; Menisci;
MeSH Terms: conditions — Osteoarthritis, Knee; Knee Injuries

STUDY DESIGN:
Intervention Model Description: It was a randomized controlled trial with two groups. One group was experimental while other group was active control group.
Who Masked: Participant
Masking Description: The participants were randomly allocated to both groups and they did not know which one was experimental or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A was given hot pack at knee joint for 10-15min. Then the Mulligan's Squeeze Technique was applied. The patient in supine lying. The therapist placed thumb on joint line tenderness of knee. With the other thumb, the therapist reinforced the first thumb. The patient was asked to slowly flex knee. The therapist maintaining the thumb contact, applied the force centrally. The force was increased progressively as the knee moved towards full range of available flexion. At the end range, the therapist assisted the tibia to move towards more flexion with ulnar border of their hand. This position was maintained for a few seconds and the overpressure was applied. Then patient was asked to perform knee extension. As the knee moved towards extension the force applied from both thumbs was progressively reduced. At maximal extension, no force was applied. This was repeated 10 times in each set with total 3 sets. After this stretching and strengthening exercises were performed by patient.
  Interventions: Other: Mulligan's Squeeze Technique - manual therapy; Other: Conventional Physiotherapy
- Group B (Active Comparator): Group B was given hot pack at knee joint for 10-15min. Then they were asked to perform stretching and strengthening exercises of the knee with at least 10 repetitions in each set and a total two sets in a day.
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Mulligan's Squeeze Technique - manual therapy — This technique was introduced by Brian R. Mulligan. In this technique the therapist places thumb along the tender joint margin and applies force centrally. The patient actively flexes knee and therapist progressively enhances force and at end applies overpressure. This force is decreased as knee moves towards extension. This method helps to maintain the meniscus in its normal position and corrects the derangement of meniscus.
  Arms: Group A
Other: Conventional Physiotherapy — It includes stretching and strengthening exercises of muscles of the knee joint.

SUMMARY:
The objective of this study is to find out the effects of Mulligan's Squeeze technique added as a complementary treatment to the conventional physiotherapy for the management of meniscal derangement in knee osteoarthritis patients.

DETAILED DESCRIPTION:
This study was performed to determine the consequences of conventional physical therapy with and without Mulligan's Squeeze technique for meniscal derangement treatment in patients with knee osteoarthritis. This research study was a randomized controlled trial. The sample size was of 26 subjects. The subjects were nominated in accordance to the inclusion and exclusion criteria. They were equally and randomly divided into two groups. One group received Mulligan's Squeeze technique along with conventional physiotherapy exercises, with hot pack prior to the exercise session. The control group was only given conventional therapy exercises with hot pack application prior to any exercise. The treatment was given for two weeks and a total of six sessions, three sessions each week. The primary outcome measures were Numerical Pain Rating Scale (NPRS) for pain rating and goniometer to record range of knee flexion. The secondary outcome measures were Patient-specific functional scale (PSFS) and Knee-injury osteoarthritis outcome score (KOOS). The measurements were taken at baseline, at end of first week and after the second week. The data was analyzed by using IBM SPSS software version 27.

ELIGIBILITY:
Inclusion Criteria:

* • Pain during maximal knee flexion, pain when maximal extension of knee occurs

  * Both genders were taken; male and female
  * Age between 30 to 55 years
  * Tenderness along the line of joint
  * Complain or history of abnormal clicking sounds and/or popping of knee
  * If any of the mentioned special tests are positive: "Apley's compression and distraction test", the "Disco test or Thessaly's test" with almost 20° flexed position of knee, and "McMurray's test"
  * Participants who were willing to take part in the study

Exclusion Criteria:

* • Presence of any knee co-morbidities

  * Knee OA of Grade 4
  * ACL or some other knee ligament injury/tears
  * Contusion present on knee, fracture of knee
  * Knee dislocation
  * Knee instability due to any ligamentous injury
  * Constant pain or discomfort due to underlying reasons (e.g. hyper-algesia), and any other wound or ailment
  * Participant not willing to be a part of the study

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | Readings were taken at baseline, after 1st week and at end of 2nd week.
  It was used to record the level of knee pain
Goniometer | Readings were taken at baseline, after 1st week and at end of 2nd week.
  It was used to find out the range of movement of knee flexion.

SECONDARY OUTCOMES:
Patient Specific Functional Scale (PSFS) | Readings were taken at baseline, after 1st week and at end of 2nd week.
  It was used to find out the independence level and dysfunction level of patient.
Knee injury and osteoarthritis outcome score (KOOS) | Readings were taken at baseline, after 1st week and at end of 2nd week.
  It is a scale designed specifically for knee problems. It has forty-two questions that cover several aspects of the problems related to knee.

CONTACTS AND LOCATIONS:
Locations (1):
- Allied Hospital, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided